CLINICAL TRIAL: NCT00226850
Title: Using Hypnosis to Help Children Undergoing a Difficult Medical Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1HUK610
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2005-09-27 (Estimated); Status verified 2005-09

CONDITIONS: Voiding Cystourethrogram (VCUG)
MeSH Terms: interventions — Hypnosis

INTERVENTIONS:
Behavioral: hypnosis

SUMMARY:
This study examined whether a hypnosis intervention, compared to standard care, could help reduce distress and pain for children undergoing an invasive medical procedure.

ELIGIBILITY:
Inclusion Criteria:

* The child: (1) was scheduled for an upcoming VCUG ; (2) must have undergone at least one previous VCUG; (3) was at least 4 years of age at the time of the previous VCUG; (4) experienced distress during the previous VCUG; and (5) both child and participating parent were English speaking.

Exclusion Criteria:

* Not meeting any of the above criteria.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D. Butler, Ph.D., Study Director — Stanford University; David Spiegel, M.D., Principal Investigator — Stanford University; Linda D Shortliffe, M.D., Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Department of Psychiatry & Behavioral Sciences, Stanford University School of Medicine, Stanford, California
  - Lucile Packard Children's Hospital, Stanford, California

REFERENCES:
- [Result] Butler LD, Symons BK, Henderson SL, Shortliffe LD, Spiegel D. Hypnosis reduces distress and duration of an invasive medical procedure for children. Pediatrics. 2005 Jan;115(1):e77-85. doi: 10.1542/peds.2004-0818. PMID 15629969